CLINICAL TRIAL: NCT00159575
Title: Metformin Treatment Before IVF / ICSI in Non-obese Women With Polycystic Ovarian Syndrome
Brief Title: Metformin in Assisted Reproduction-MET-AR-study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow patient recruitment and expiry of study medication(aug2009)
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MET-AR study -PCOS 5; EUDRACTNR. 2004-001124-20
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic ovarian syndrome; Clinical pregnancy rate; Oligo- or anovulation
MeSH Terms: conditions — Polycystic Ovary Syndrome; Anovulation | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- M: Metformin P: Placebo (Experimental)
  Interventions: Drug: Metformin / Placebo treatment for 4 months

INTERVENTIONS:
Drug: Metformin / Placebo treatment for 4 months — M: Metformin 2000mg daily- 12-14 weeks of pretreatment + metformin 2000mg daily through conventional IVF ending on the day of pregnancy test; IE. 14 days after embryo transfer. P: Or identical placebo treatment for the same period

SUMMARY:
Aim of study: To investigate whether four months of metformin treatment before IVF (in-vitro-fertilisation) or ICSI (intra-cytoplasmic-sperm-injection) might increase clinical pregnancy rate in normal-weight (body mass index [BMI] below 28 kg/m3) in PCOS (polycystic ovarian syndrome) women.

DETAILED DESCRIPTION:
PCOS is an hormonal disease including hyperandrogenism, oligo-or anovulation and/or polycystic ovaries by ultrasound. PCOS women often suffer insulin resistance or even diabetes risk as well as a full blown metabolic disease.

These women often suffer infertility due to their lack of regular ovulations. Metformin is a well known anti-diabetic drug, and in some PCOS women metformin might decrease the hyperandrogenism, improve insulin resistance and give more regular ovulations. Thereby increase chance of pregnancy. Our hypothesis is that metformin will increase clinical pregnancy rates both spontaneously and following IVF/ICSI.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilling Rotterdam criteria for PCOS
* Infertility more than 1 year
* First or second cycle of IVF/ICSI treatment
* Age below 38 years at inclusion
* BMI below 28 kg/m3 at inclusion
* Willing to be randomised to 4 months metformin or placebo
* Signed written informed consent

Exclusion Criteria:

* Not suitable for starting dose 112.5 IE
* Basal FSH above 10 IU/L
* Known renal disease or s-creatinine above 110 umol/L
* Known liver disease or s-ALAT above 80 IU/L
* Known alcoholism or drug abuse
* Known diabetes mellitus or fasting plasma glucose above 7 mmol/L
* Corticosteroid treatment (oral)
* Treatment with cimetidine, anticoagulants, erythromycin or other macrolides
* Hyperprolactinemia (PRL above 700 mIU/L)
* Abnormal thyroid function tests
* Known congenital adrenal hyperplasia
* Androgen secreting tumours
* Cushing syndrome
* Metformin treatment within the last one month prior to screening
* Unfit to participate for any other reason

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2005-03; Primary Completion 2009-08 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
To investigate whether four months of Metformin treatment before IVF (in-vitro-fertilisation) or ICSI (intra-cytoplasmic sperm injection) will increase clinical pregnancy rate in normal weight PCOS-women | Vaginal ultrasound in pregnancy week 7

SECONDARY OUTCOMES:
Spontaneous pregnancy rates during the pretreatment period, Spontaneous abortion rates (I or II trim.abortions), Live birth rates, | Vaginal ultrasound in pregnancy week 7
Number of oocytes collected, Embryo quality, Number of days of gonadotrophin treatment, Dose of gonadotrophin, total per cycle and daily, s-estradiol on day of hCG-administration, Occurrence of ovarian hyperstimulation syndrome (OHSS) | All data evaluated at study end, from september 2009 onwards

CONTACTS AND LOCATIONS:
Overall Officials: Sven Carlsen, MD,PhD, Study Chair — St Olavs Hospital- Endocrinological section
Locations (2):
- Norway (2):
  - Sigrun Kjøtrød, Trondheim
  - Fertility UNit- -St Olavs Hospital, Trondheim

REFERENCES:
- [Result] Kjotrod SB, Carlsen SM, Rasmussen PE, Holst-Larsen T, Mellembakken J, Thurin-Kjellberg A, Haapaniemikouru K, Morin-Papunen L, Humaidan P, Sunde A, von During V. Use of metformin before and during assisted reproductive technology in non-obese young infertile women with polycystic ovary syndrome: a prospective, randomized, double-blind, multi-centre study. Hum Reprod. 2011 Aug;26(8):2045-53. doi: 10.1093/humrep/der154. Epub 2011 May 23. PMID 21606131
- [Derived] Tso LO, Costello MF, Albuquerque LET, Andriolo RB, Macedo CR. Metformin treatment before and during IVF or ICSI in women with polycystic ovary syndrome. Cochrane Database Syst Rev. 2020 Dec 21;12(12):CD006105. doi: 10.1002/14651858.CD006105.pub4. PMID 33347618